CLINICAL TRIAL: NCT04330066
Title: Impact of Endometrial Compaction in Euploid Frozen Embryo Transfers: a Prospective Observational Pilot Study
Brief Title: Impact of Endometrial Compaction in Euploid Frozen Embryo Transfers
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Boston IVF (Other)
Responsible Party: Sponsor
Other Study IDs: 2020P000191
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Infertility, Female
Keywords: endometrial compaction; frozen embryo transfer; euploid embryo; ultrasound
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exogenous hormone replacement thaw cycle: Participants in this group will follow Boston IVF's standard exogenous hormone replacement protocol. Participants will take Estrace 3mg twice daily by mouth for endometrial preparation. After 16-18 days of Estrace, endometrial thickness will be measured by transvaginal ultrasound but medication and ultrasounds will be continued until the endometrial lining is ≥ 7 mm. Once the final endometrial lining is ≥ 7 mm (T1), the doctor of record will start the participant the following day with intramuscular progesterone daily or intramuscular progesterone every 3 days with daily vaginal progesterone. Frozen embryo transfers would occur on the sixth day of progesterone.
  Interventions: Diagnostic Test: Abdominal ultrasound measurement of the endometrial lining
- Natural thaw cycle: Participants in this group will follow Boston IVF's standard natural thaw cycle protocol. Participants will be coming for blood and transvaginal ultrasound monitoring around day 11 of the participants cycle. Once the participant has a final measurement of the endometrial lining ≥ 7 mm (T1), a 17mm ovarian follicle, and a progesterone < 1.2 ng/mL, the doctor of record will schedule the patient to receive a trigger injection to induce ovulation followed by an embryo transfer 6-7 days later. Participants may be started on vaginal progesterone 4 days after the trigger injection for added supplementation per the doctor of record.
  Interventions: Diagnostic Test: Abdominal ultrasound measurement of the endometrial lining

INTERVENTIONS:
Diagnostic Test: Abdominal ultrasound measurement of the endometrial lining — On the day of the participants frozen embryo transfer, an endometrial thickness measurement (T2) will obtained from an abdominal ultrasound during the embryo transfer.

SUMMARY:
The purpose of this pilot study is to evaluate whether a decrease in endometrial thickness (compaction) prior to progesterone exposure (endogenous or exogenous) to the day before a single frozen embryo transfer has an impact on the clinical pregnancy rate with euploid embryos in exogenous hormone and modified natural thaw cycles. Information derived from this study may give insight on ways to improve pregnancy rates in cryo-thaw cycles.

DETAILED DESCRIPTION:
Methods: Study participation will not influence any element of IVF treatment and all participants will be receiving the standard of care at Boston IVF. Potential participants will be identified by a member of the research team, who will review the appointment log and medical records to ensure eligibility. Eligible participants interested in participating in the study will have an abdominal ultrasound endometrial thickness measurement on the day of the participants embryo transfer (T2). This abdominal ultrasound is part of routine clinical care necessary for the embryo transfer. The eligible participant will provide verbal consent to a member of the research team prior to the ultrasound. Baseline demographic data will be obtained from the electronic medical record including: age, race, education level, partner status, height, weight, gravidity, and parity.

Two groups of thaw cycles will be included: (1) exogenous hormone replacement thaw cycles and (2) modified natural thaw cycle. Both groups will follow the standard of care for cycle preparation at Boston IVF. Ultrasound measurements of the endometrial lining (T1) will only be used if they were within 1 day of the initiation of progesterone (group 1) or ovulation trigger injection (group 2). At T1, multiple endometrial lining measurements will be made per standard protocol, but only the optimal image and measurement will be saved. At T2, only a single endometrial thickness measurement will be measured by the sonographer and will be recorded on a study log. Images should include a longitudinal view of the endometrium and cervix. Measurements from the T2 ultrasound will be blinded from the participant and they will not be used to make any clinical decisions. Both groups will have a comparison of the difference in endometrial thickness measurement between T1 and T2.

Sample Size Justification: Given the limited data on this specific topic, the study will be an observational pilot study. Given the available resources, the researchers will aim to have 100 participants per cycle preparation group, for a total of 200 participants.

Data Analysis: Descriptive data will be presented as the proportion, mean with standard deviation, or median with interquartile range. Comparisons will be made using the chi-square or Fisher's exact test for categorical variables and parametric or non-parametric tests for continuous variables based on data distribution. Logistic regression analysis will be performed for multivariate analysis. All data will be analyzed with SAS 9.4 (SAS Institute Inc., Cary, NC, USA). All tests will be two sided and a P value < 0.05 will be required to confer significance.

ELIGIBILITY:
Inclusion Criteria:

* Single euploid frozen embryo transfer
* ≥ 7 mm endometrial lining on transvaginal ultrasound
* 1st or 2nd frozen embryo transfer

Exclusion Criteria:

* Obesity with body mass index > 40
* Underweight with body mass index < 18.5
* Utilization of a gestational carrier
* History of recurrent pregnancy loss (≥ 2 spontaneous abortions)
* Uterine factors (history of uterine adhesions, uterine surgery, fibroids, polyps)
* History of an endometrial receptivity assay (ERA) biopsy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants that are having a single frozen embryo transfer with a euploid embryo.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | through study completion, an average of 1 year
  defined as confirmation of gestational sac with fetal heart beat on ultrasound between 6 - 9 weeks gestation

SECONDARY OUTCOMES:
Biochemical pregnancy rate | through study completion, an average of 1 year
  defined as positive beta-hCG but no gestational sac visualized
Live birth rate | through study completion, an average of 1 year
  defined as delivery > 23 weeks gestation
Miscarriage rate | through study completion, an average of 1 year
  defined as the loss of a pregnancy prior to 12 weeks per total number of pregnancies

CONTACTS AND LOCATIONS:
Overall Officials: Alan Penzias, MD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah JS, Vaughan DA, Dodge LE, Leung A, Korkidakis A, Sakkas D, Ryley DA, Penzias AS, Toth TL. Endometrial compaction does not predict live birth in single euploid frozen embryo transfers: a prospective study. Hum Reprod. 2022 May 3;37(5):980-987. doi: 10.1093/humrep/deac060. PMID 35357436